CLINICAL TRIAL: NCT05131139
Title: Enhance Study: A Prospective, Multicenter Evaluation of Accuracy and Safety of the Eversense CGM System With Enhanced Features
Brief Title: Enhance Study: Evaluation of Accuracy and Safety of the Eversense CGM System With Enhanced Features
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0041
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Continuous Glucose Monitoring Device (Experimental): Eversense 524 CGM System and ROME CGM System.
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Eversense 524 CGM System and ROME CGM System.

SUMMARY:
A Prospective, Multicenter Evaluation of Accuracy and Safety of the Eversense CGM System with Enhanced Features. The purpose of this clinical investigation is to evaluate the accuracy of the Eversense 524 Continuous Glucose Monitoring System (Eversense 524 CGM System) and ROME CGM System with next generation feature enhancements compared to reference glucose measurements in adults 18 years of age and older with diabetes. The investigation will also evaluate safety of the Eversense 524 CGM System and ROME CGM System usage. Additionally, the safety and accuracy of the Eversense 524 CGM System will be evaluated in the pediatric population ages 14-17 with Type 1 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following inclusion criteria will be included in this study:

1. Subjects ≥14 years of age
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year for adults 18 years and older
3. Clinically confirmed diagnosis of type I diabetes mellitus for ≥1 year for adolescents 14 -17 years old
4. Subject has signed an informed consent or assent form and parent/guardian has signed an informed consent, as applicable, and subject is willing to comply with protocol requirements.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria at the time of screening will be excluded from this study:

1. History of unexplained severe hypoglycemia in the previous 6 months. Severe hypoglycemia is defined as hypoglycemia resulting in loss of consciousness or seizure.
2. History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months.
3. Subjects with gastroparesis.
4. Female subjects of childbearing capacity (defined as of child bearing age and as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study.
5. A condition preventing or complicating the placement, operation, or removal of the sensor or wearing of transmitter, including upper extremity deformities or skin condition.
6. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke in the past 6 months; uncontrolled hypertension (systolic>160 mm Hg or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign PACs and PVCs allowed). Subjects with asymptomatic coronary artery disease (e.g., CABG, stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from Cardiologist documented.
7. Hematocrit <38% or >60% at screening
8. History of hepatitis B, hepatitis C, or HIV
9. Current treatment for a seizure disorder unless written clearance by neurologist to participate in study.
10. History of adrenal insufficiency
11. Currently receiving (or likely to need during the study period): immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin); topical glucocorticoids over sensor site only; antibiotic for chronic infection (e.g., osteomyelitis, endocarditis)
12. For subjects inserted with the ROME CGM System: A condition requiring or likely to require magnetic resonance imaging (MRI)
13. Known topical or local anesthetic allergy
14. Known allergy to glucocorticoids
15. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study. Conditions include but are not limited to psychiatric conditions, known current or recent alcohol abuse or drug abuse by subject history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
16. Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
17. The presence of any other active implanted device (as defined further in protocol)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Objective: To determine accuracy of the Eversense 524 CGM System and ROME CGM System. | 365 days
  The effectiveness measure will be mean absolute relative difference (MARD) for paired sensor and reference measurements through 365 days post-insertion for reference glucose values from 40-400 mg/dL. Effectiveness measures will be evaluated descriptively.
Safety Objective: To demonstrate safety of the Eversense 524 CGM System and ROME CGM System. | 365 days
  Incidence of device-related or sensor insertion/removal procedure-related serious adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - AMCR Institute Inc., Escondido, California
  - Rocky Mountain Diabetes Center, LLC. (RMDC), Idaho Falls, Idaho
  - Clinical Trials of Texas, LLC. (CTT), San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No